CLINICAL TRIAL: NCT03326401
Title: The Evaluation of Nutrition Status in Persons With Age-Related Macular Degeneration
Brief Title: The Potential Role of Dietary Antioxidant Capacity on Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, F. Gülhan Samur, Associate Professor, Hacettepe University
Other Study IDs: GO 15/628
Record Dates: First submitted 2017-10-19; First posted 2017-10-31 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Age Related Macular Degeneration
Keywords: dietary total antioxidant activity; nutritional status; macular degeneration; glycemic load; glycemic index; nutrient intake
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case (AMD group): Case group including 100 patients diagnosed with age-related macular degeneration (50 women, 50 men).Demographic data and dietary intake of different food groups were assessed by a standardized interviewer-assisted questionaire with the method of face-to-face interview. The body weight of the individuals were measured with a calibrated electronic scale,anthropometric measurements were measured by the researcher. Participants' dietary intake was assessed using food frequency questionaire (FFQ). The FFQ included 65 food items traditionally consumed in Turkey. Foods were classified into the following food categories: milk and dairy products, meat and meat products, fruits, vegetables, breads and cereals, beverages, and desserts.
- Control (Non-AMD group): Case group including 100 patients not diagnosed with age-related macular degeneration (50 women, 50 men).Demographic data and dietary intake of different food groups were assessed by a standardized interviewer-assisted questionaire with the method of face-to-face interview. The questionaire form, prepared to determine socio-demographic features of individuals participating in the research, was applied by the research with the method of face-to-face interview. The body weight of the individuals were measured with a calibrated electronic scale,anthropometric measurements were measured by the researcher. Participants' dietary intake was assessed using food frequency questionaire (FFQ). The FFQ included 65 food items traditionally consumed in Turkey. Foods were classified into the following food categories: milk and dairy products, meat and meat products, fruits, vegetables, breads and cereals, beverages, and desserts.

SUMMARY:
Including eye health, nutrition plays a vital role for the sustainability of individuals health life. There is an increasing global concern about the issues related with eye health. In 2010, in order to take attention to these issues, World Health Organization (WHO) defined the main reasons of vision disorders as refraction defects of eye diseases (43 %), cataract (33 %), glaucoma (2 %), age-related macular degeneration (AMD) (1 %), diabetic retinopathy (1 %) and undetermined natural reasons (18 %). This report also stated the three biggest reasons of blindness as cataract (51 %), glaucoma (8 %) and AMD (5 %).

AMD is a multi-factorial disease in which the genetic predisposition plays important role with environmental factors and metabolic conditions, except for age. Especially cigarette is the secondary important risk factor for dry-type AMD. In the Age Related Eye Disease Study (AREDS), it was stated that AMD prevalence is higher in white races, compared with races which are not white. At the same time, AREDS searched the effect of diet supplements on the progression of AMD disease. In terms of the patients followed for six years, it was reported that the formulation C and E vitamins, beta carotene and zinc decreased the progression risk of AMD from middle levels to advanced levels by 34 %. In AREDS-2 study completed in 2012, it was shown that the extraction of beta carotene from the formulation and the decrease of zinc did not affect the progression rate of the disease. In the group using beta carotene, including persons who were used to smoke but gave up at least one year ago, the rate of becoming lung cancer was observed as substantially high. Moreover, the use of lutein and zeaxanthin instead of beta carotene in the formula did not increase the risk of lung cancer. In addition, it was shown that omega-3 fatty acids did not decrease risk progression.

In current data, the effect of the intake of carotenoid and antioxidant increased with diet on AMD is not coherent. Likewise, the epidemiological evidences about the relation between diet fat intake and AMD are contradictory. The consumption of fatty fish is related with increased poly-unsaturated fatty acid intake and decreases the risk of AMD. However, it was reported the high rate of total fat intake in other studies as risk factor for AMD. In another study, there was not any important relation found between diet fat intake and AMD occurrence after the correction of other variables. In the interventional AREDS-2 study, it was reported that the additional intake of long-chain omega-3 poly-unsaturated fatty acids did not have any beneficial effect.

The pathophysiological mechanism responsible from the possible relation between obesity and AMD is not clearly known. There are various hypotheses about how obesity causes AMD. In the first hypothesis, obesity can cause AMD after obesity increases systematic oxidative stress. In the second hypothesis, obesity can play a role in AMD pathophysiology as the cause of hyperleptinemia. The studies also prescribed that inflammation could play a role in the progression of AMD and also showed that plasma fibrinogen and other inflammation indicators could be related with late AMD. In Pathologies Oculaires Liées à l'Age (POLA) study made with the participation of many Europeans, it was observed that the progression of late AMD increased by two times in obese individuals and in early AMD, obesity did not affect the progression of disease. In the treatment of this disease which have age-related progression, proper nutrition, vitamin/mineral/supplement usage and the development of precautionary strategies play an important role.

When compared with Body Mass Index (BMI), it was found that the measure of abdominal obesity (waist/hip rate and waist circumference) was the better determinant of chronic diseases such as diabetics and cardiovascular disease. Some evidences in the United States of America indicated that the relation between waist/hip rate and AMD gave stronger results when compared with the relation between BMI and AMD. For middle age cohort, after six years of follow-up, a group of researchers reported that the decrease of waist/hip rate also decreased the risk of AMD and the results were the same for waist circumference, even if the evidences were weak. In another study, it was reported that the increase of waist/hip rate or waist circumference also increased the progression of AMD.

This study was planned with the aim of determining the occurrence of AMD by evaluating dietary total antioxidant capacity, diet components and some anthropometric measures of individuals having age related macular degeneration (AMD). In the study, the possible effect of nutrition on the occurrence of disease was evaluated by comparing healthy individuals with dietary total antioxidant capacity and some anthropometric measures of individuals with AMD.

DETAILED DESCRIPTION:
While being benefited from the results of previous studies, the sample size of the research was type 1 error performance α=0.05 and type 2 error performance β=0.20. The power of the test was taken as 1-β=0.80 and the power analysis was statistically made with NCCS PAS 11 program. 200 individuals voluntarily participated into the study as control group, including 100 patients diagnosed with AMD (50 women, 50 men) and 100 patients not diagnosed as AMD (50 women, 50 men).

Sociodemographic Variables The questionnaire form, prepared to determine socio-demographic features of individuals participating in the research, was applied by the research with the method of face-to-face interview. The socio-demographic features of individuals (gender, age, occupation, educational status, health conditions), use of cigarettes and drugs was questioned.

Anthropometric Variables The body weight of the individuals were measured with a calibrated electronic scale, which could measure even 0.1 kg, while the individuals were hungry, in light clothes and their shoes were taken off. The body lengths were measured by the researcher with the tape measure while they were standing upright in Frankfurt plane position (ear canal and lower margin of orbit in the same horizontal plane, facing forward). BMI was calculated with the formula [body weight (kg)/body length (m2)]. BMI evaluation was made while the classification developed by World Health Organization (WHO) was taken as a basis (13). According to this classification; (BMI<18.5 kg/m2 thin, 18.5< 24.9 kg/m2 normal, 25.0-29.9 kg/m2 overweight and ≥30 kg/m2 obese. The waist circumference of the individuals was measured with tape measure by founding the midpoint between the lowest rib and umbilicus. The relation between waist circumference and chronic diseases is as follows: If the waist circumference is ≥88 cm for women and ≥102 cm for men, it is shown as high risk. The hip circumference of the individuals was measured with a tape measure from the highest point by standing the left side of the individuals. If the waist/hip rate is over 0.85 for women and over 0.90 for men, the risk of chronic diseases increases.

Assesment of dietary intake and diet total antioxidant capacity Participants' dietary intake was assessed using food frequency questionnaire (FFQ). The FFQ included 65 food items traditionally consumed in Turkey. Foods were classified into the following food categories: milk and dairy products, meat and meat products, fruits, vegetables, breads and cereals, beverages, and desserts. Intake frequencies for the food items consisted of eight categories ranging from never/once a month to more than one per day. Trained interviewers asked participants how often they had consumed one portion of each food item in generally. To compute the total amount of food intake per day, the reported frequency of consumption for each food item was multiplied by the portion size and then total food intake was converted to nutrient intake based on the food's nutrient profile. Standardized food recipes for Turkey and Nutrition Information System (BEBIS) program which is a food composition database for nutrient estimation were used to determine average daily energy and nutrient intake for each participant. These values were compared with the recommended daily allowance values to determine the energy and nutrient requirement meeting status and the requirement meeting percentages were calculated.

By using food intake frequency amounts, dietary total antioxidant capacity was tried to be determined approximately with the use of data obtained from a large-scale study made by Carlsen for developing a database including total antioxidant component of essential nutrients. The antioxidant amount in 100 g food given for each nutrient group in the related resource was used as standard antioxidant activity value in this study and the approximate antioxidant activity values of the grouped food intake amounts of individuals were calculated.

Statistical Analysis In the statistical evaluation of data obtained from the study, Statistical Package for Social Science (SPSS) 22.0 program was used. For the data obtained from the measures of individuals participating in the study, average, standard deviation and the lowest and the highest values were calculated. The distribution of data determined with numbers was given with number-percentage tables. While evaluating constant data, it was determined with Kolmogorov Smirnov test whether there was normal distribution or not. The data of individuals having normal distribution were analyzed with parametric statistical tests and the data of individuals not having normal distribution were analyzed with non-parametric statistical tests. Odds ratios (OR) and 95% confidence intervals (CI) were calculated by univariate logistic regression analysis separately for food group, BMI, and adjusted age, gender before combined in multivariate logistic regression. Logistic regression analysis was performed to determine risk factors for AMD using odds ratio estimates with 95% confidence intervals. Furthermore, a stepwise multivariate regression analysis was performed, with p value less than 0.05 being required for entering the model and remaining there.

ELIGIBILITY:
Inclusion Criteria:

* Subject older than 50 years old
* Clinical diagnosis of Age-Related Macular Degeneration Disease (Both Dry and Wet type)

Exclusion Criteria:

* Subject complying with a special diet
* History of cardiovascular disease
* History of eye surgery
* Subject younger than 50 years old

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 200 individuals voluntarily participated into the study including 100 patients diagnosed with AMD (50 women, 50 men) and 100 patients not diagnosed as AMD (50 women, 50 men) as control group.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2016-02-20 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | up to 20 weeks
  It will calculate by researcher with BMI formula: kg/m^2
Dietary total antioxidant capacity of participants | up to 20 weeks
  3 day food record of participants will be taken and evaluated by researcher. Nutrition information System (BeBİS) software will be used for calculate daily consumption of nutrients.

CONTACTS AND LOCATIONS:
Overall Officials: F.Gülhan Samur, Ass. Prof., Principal Investigator — Hacettepe University; Sibel Kadayıfçılar, Prof., Study Chair — Hacettepe University; Sedat Arslan, RA, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University Hospital Department of Ophthalmology Polyclinic, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol will be shared with other researches in one year.

REFERENCES:
- [Result] Schaumberg DA, Christen WG, Hankinson SE, Glynn RJ. Body mass index and the incidence of visually significant age-related maculopathy in men. Arch Ophthalmol. 2001 Sep;119(9):1259-65. doi: 10.1001/archopht.119.9.1259. PMID 11545630
- [Result] Klein BE, Klein R, Lee KE, Jensen SC. Measures of obesity and age-related eye diseases. Ophthalmic Epidemiol. 2001 Sep;8(4):251-62. doi: 10.1076/opep.8.4.251.1612. PMID 11471093
- [Result] Clemons TE, Milton RC, Klein R, Seddon JM, Ferris FL 3rd; Age-Related Eye Disease Study Research Group. Risk factors for the incidence of Advanced Age-Related Macular Degeneration in the Age-Related Eye Disease Study (AREDS) AREDS report no. 19. Ophthalmology. 2005 Apr;112(4):533-9. doi: 10.1016/j.ophtha.2004.10.047. PMID 15808240
- [Result] Defay R, Delcourt C, Ranvier M, Lacroux A, Papoz L. Relationships between physical activity, obesity and diabetes mellitus in a French elderly population: the POLA study. Pathologies Oculaires liees a l' Age. Int J Obes Relat Metab Disord. 2001 Apr;25(4):512-8. doi: 10.1038/sj.ijo.0801570. PMID 11319655
- [Result] Smith W, Assink J, Klein R, Mitchell P, Klaver CC, Klein BE, Hofman A, Jensen S, Wang JJ, de Jong PT. Risk factors for age-related macular degeneration: Pooled findings from three continents. Ophthalmology. 2001 Apr;108(4):697-704. doi: 10.1016/s0161-6420(00)00580-7. PMID 11297486
- [Result] Seddon JM, Cote J, Davis N, Rosner B. Progression of age-related macular degeneration: association with body mass index, waist circumference, and waist-hip ratio. Arch Ophthalmol. 2003 Jun;121(6):785-92. doi: 10.1001/archopht.121.6.785. PMID 12796248
- [Result] Cho E, Seddon JM, Rosner B, Willett WC, Hankinson SE. Prospective study of intake of fruits, vegetables, vitamins, and carotenoids and risk of age-related maculopathy. Arch Ophthalmol. 2004 Jun;122(6):883-92. doi: 10.1001/archopht.122.6.883. PMID 15197064
- See also: who bmi classification — http://www.euro.who.int/en/health-topics/disease-prevention/nutrition/a-healthy-lifestyle/body-mass-index-bmi
- See also: nutrition information system — http://bebis.com.tr/